CLINICAL TRIAL: NCT06916403
Title: A Two-part Study to Access the Safety and Efficacy of Ketamine Intravenous Infusions in the Treatment of Fibromyalgia
Brief Title: Safety and Efficacy of Ketamine Intravenous Infusions in the Treatment of Fibromyalgia
Status: Active, not recruiting | Type: Observational
Sponsor: Wilderman Medical Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: WMC003
Record Dates: First submitted 2025-03-24; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Intravenous Ketamine Infusions; Chronic Pain; Neuropathic Pain; Dissociative State; Depression; Pain Relief
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Neuralgia; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective Study Group: A total of approximately 30 patients diagnosed with fibromyalgia will be selected for participation in the study, all of whom will be treated with one IV ketamine infusion for pain relief according to their regular schedule of IV ketamine infusions.
  Each patient will be evaluated at baseline (prior to ketamine infusion), 40 minutes post-infusion, and at follow up visits.
  Interventions: Drug: Intravenous Ketamine Infusions
- Retrospective Study group: A total of approximately 20 patients will be selected for participation in the study, all of whom were treated with IV ketamine infusions. Information regarding clinically relevant outcomes will be obtained from chart reviews from patients who meet the eligibility criteria.
  The patient's response to treatment will be assessed.
  Interventions: Drug: Intravenous Ketamine Infusions

INTERVENTIONS:
Drug: Intravenous Ketamine Infusions — Ketamine will be slowly infused with the routine target dose 1.5-2 mg/kg over 3-4 hours.

SUMMARY:
Previous studies of intravenous ketamine, which is a non-competitive N-methyl-D aspartate receptor antagonist, for fibromyalgia pain relief are limited to three studies. Two studies have focused on short-term pain relief of intravenous ketamine by measuring the patients' pain levels immediately before and after the infusion. Currently, existing studies used short-term infusions (30-40 minutes) of sub-anesthetic doses of ketamine for pain relief in fibromyalgia patients, whereas the Consensus Guidelines on the Use of Intravenous Ketamine Infusions for Chronic Pain from the American Society of Regional Anesthesia and Pain Medicine, the American Academy of Pain Medicine, and the American Society of Anesthesiologists recommend infusing IV ketamine for at least two hours and a minimal total dose of 80 mg.

The rationale of this study is to expand on the existing data of safety and efficacy of intravenous ketamine to relieve fibromyalgia pain. Specifically, this investigation will add data to fill the existing gap regarding the short- and long-term pain relief in the treatment of fibromyalgia with intravenous ketamine infusions. The study will also attempt to determine safety and tolerability. In addition, the characteristics of treatment responders versus non-responders will be assessed in an effort to determine whether specific characteristics can be used to predict treatment response in this group of patients.

DETAILED DESCRIPTION:
This study consists of two parts. The first part is a single-centre, retrospective chart review to analyze and summarize the investigators' experience with intravenous ketamine infusions in the treatment of patients with fibromyalgia who received at least four infusions for pain management. For the second part, patients who already received at least three intravenous ketamine infusions (for optimal dose determination) will be enrolled in an open single-group prospective study to receive one intravenous ketamine treatment. In this prospective study, the investigators will evaluate infusion effectiveness, safety, and tolerability as well as the influence of patients' demographic and medical characteristics, including depression status and ketamine dissociation symptoms, on the treatment outcome.

This two-part study aims to evaluate whether intravenous ketamine is effective in reducing pain in patients diagnosed with fibromyalgia. To achieve this goal, the study will assess the effect of intravenous ketamine infusions on short- and long-term pain relief. The study will also evaluate the safety and tolerability of ketamine infusions in fibromyalgia patients and factors that may have an impact on the treatment outcome.

ELIGIBILITY:
Inclusion criteria:

To be included in Part 1 of the study, patients must fulfil the following criteria:

* Given written consent to permit Wilderman Medical Clinic investigators to use their medical and demographic information in research studies.
* Male or female >18 years of age
* Having been diagnosed with fibromyalgia
* Received at least 4 IV ketamine infusion(s)
* Made at least one rating of pain (NRS) immediately before the intervention and one after the intervention
* Had follow-up data recorded on the follow-up visit: percentage and duration of pain relief

To be included in Part 2 of the study, patients must fulfil the following criteria:

* Male or female >18 years of age
* Given the written Informed Consent Form to participate in the study
* Having been diagnosed with fibromyalgia
* Having been prescribed IV ketamine infusions treatment
* Passed safety screening for ketamine infusions
* Had at least 3 IV ketamine infusions for dose optimization
* Willingness and ability to comply with the study procedure and the ability to follow verbal and written instructions

Exclusion Criteria:

Patients will be excluded from Part 1 of the study if they meet any of the following criteria:

* Age less than 18 years old
* Absence of signed Informed Consent Form
* Patients who received less than 4 IV ketamine infusion(s)
* Insufficient information to conduct analysis (e.g. absence of pain ratings or follow up measurements)

Patients will be excluded from the Part II of the study if they meet any of the following criteria:

* Age less than 18 years old
* Absence of signed Informed Consent Form
* Received less than 3 IV ketamine infusions
* Have any contradictions to the administration of intravenous ketamine (known allergy to ketamine or fail to pass Ketamine treatment screening)
* Diagnosis of dementia or other cognitive impairments
* Any clinically significant acute or chronic medical condition that in the judgment of Investigator may preclude the use of intravenous ketamine or compromise patient safety, limit patient's ability to complete the study, and/or compromise the objectives of the study.
* Participation in any other clinical study within 3 months prior to screening and during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from Wilderman Medical Clinic, a chronic pain clinic located in Thornhill, Ontario. The clinic consists of state-of-the-art out-patient facilities, an interdisciplinary team and nursing support.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) | Baseline visit: immediately before IV ketamine infusion
  The NRS is a standardized, one-dimensional measure of pain intensity. The pain intensity is rated by the participant using a scale from 0-10; 0 being the least (no pain) to 10 (worst pain imaginable).
Numeric Rating Scale (NRS) | Baseline visit: immediately after the IV ketamine infusion
  The NRS is a standardized, one-dimensional measure of pain intensity. The pain intensity is rated by the participant using a scale from 0-10; 0 being the least (no pain) to 10 (worst pain imaginable).
Numeric Rating Scale (NRS) | Follow-up visits at 1, 2, 3, and 4 weeks after the IV ketamine infusion
  The NRS is a standardized, one-dimensional measure of pain intensity. The pain intensity is rated by the participant using a scale from 0-10; 0 being the least (no pain) to 10 (worst pain imaginable).
Integral of pain relief | Follow-up visits at 1, 2, 3, and 4 weeks after the IV ketamine infusion
  IPR is a multidimensional measure combining the duration of patients' pain relief (in days) and the percentage of pain relief that they had experienced. IPR seeks to tap into a fuller picture of the patients' pain relief, since it not only measures current pain levels, but patients' experience of pain, both in duration and percentage of relief, over a longer period of time. The scale has no restrictions, beginning at 0 (no treatment effect). Therefore, the higher the IPR value, the more effective the treatment was at reducing pain

SECONDARY OUTCOMES:
The Clinician-Administered Dissociative States Scale (CADSS) | Baseline visit: immediately before IV ketamine infusion
  The CADSS is a 27-item scale with 19 subject-rated items and 8 items scored by an observer. The subjective component consists of 19 items which are administered by a clinician who begins each question with the phrase "at this time" and then reads the item to the subject. The subject then endorses one of a range of possible responses: 0 = not at all, 1 = slightly, 2 = moderately, 3 = considerably, 4 = extremely. The subject's response on these 0 to 4 scales is recorded and the clinician moves on to the next item. Three non-empirically derived subscales for the CADSS have been proposed: amnesia (two items), depersonalization (five items), and derealization (12 items).
The Clinician-Administered Dissociative States Scale (CADSS) | Baseline visit: 40 minutes after the IV ketamine infusion
  The CADSS is a 27-item scale with 19 subject-rated items and 8 items scored by an observer. The subjective component consists of 19 items which are administered by a clinician who begins each question with the phrase "at this time" and then reads the item to the subject. The subject then endorses one of a range of possible responses: 0 = not at all, 1 = slightly, 2 = moderately, 3 = considerably, 4 = extremely. The subject's response on these 0 to 4 scales is recorded and the clinician moves on to the next item. Three non-empirically derived subscales for the CADSS have been proposed: amnesia (two items), depersonalization (five items), and derealization (12 items).
Patient Health Questionnaire (PHQ-9) | Baseline visit: before IV ketamine infusion
  PHQ-9 is endorsed by the National Institute for Health and Clinical Excellence for use in primary care in measuring baseline depression severity and responsiveness to treatment. The 9 items on the PHQ-9 consist of the 9 criteria on which the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) depressive disorder diagnoses are based. A 4-point scale indicates a degree of severity; items are rated from 0 (not at all) to 3 (nearly every day).
Patient Health Questionnaire (PHQ-9) | Follow-up visits at 1, 2, 3, and 4 weeks after the IV ketamine infusion
  PHQ-9 is endorsed by the National Institute for Health and Clinical Excellence for use in primary care in measuring baseline depression severity and responsiveness to treatment. The 9 items on the PHQ-9 consist of the 9 criteria on which the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) depressive disorder diagnoses are based. A 4-point scale indicates a degree of severity; items are rated from 0 (not at all) to 3 (nearly every day).
Self-completed Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) | Baseline visit: before IV ketamine infusion
  The LANSS is a simple and valid 7-item tool for identifying patients whose pain is dominated by neuropathic mechanisms. Each item is a binary response (yes or no) to the presence of symptoms (5 items) or clinical signs (2 items). S-LANSS is a modified version of the LANSS pain scale to make it capable of self-completion.
Self-completed Leeds Assessment of Neuropathic Symptoms and Signs (S-LANSS) | Follow-up visits at 1, 2, 3, and 4 weeks after the IV ketamine infusion
  The LANSS is a simple and valid 7-item tool for identifying patients whose pain is dominated by neuropathic mechanisms. Each item is a binary response (yes or no) to the presence of symptoms (5 items) or clinical signs (2 items). S-LANSS is a modified version of the LANSS pain scale to make it capable of self-completion.
Fibromyalgia Impact Questionnaire, Revised (FIQR) | Baseline visit: before IV ketamine infusion
  The Fibromyalgia Impact Questionnaire (FIQ) is a commonly used instrument in the evaluation of fibromyalgia patients. The revised FIQ has 21 individual questions. All questions are based on an 11-point numeric rating scale of 0 to 10, with 10 being 'worst'. All questions are framed in the context of the past 7 days. The FIQR is divided into three linked sets of domains: (a) 'function' (contains 9 questions), (b) 'overall impact' (contains 2 questions), and (c) 'symptoms' (contains 10 questions). The FIQR is an updated version of the FIQ that has good psychometric properties, can be completed in less than 2 minutes and is easy to score.
Fibromyalgia Impact Questionnaire, Revised (FIQR) | Follow-up visits at 1, 2, 3, and 4 weeks after the IV ketamine infusion
  The Fibromyalgia Impact Questionnaire (FIQ) is a commonly used instrument in the evaluation of fibromyalgia patients. The revised FIQ has 21 individual questions. All questions are based on an 11-point numeric rating scale of 0 to 10, with 10 being 'worst'. All questions are framed in the context of the past 7 days. The FIQR is divided into three linked sets of domains: (a) 'function' (contains 9 questions), (b) 'overall impact' (contains 2 questions), and (c) 'symptoms' (contains 10 questions). The FIQR is an updated version of the FIQ that has good psychometric properties, can be completed in less than 2 minutes and is easy to score.
Patients Global Impression of Change (PGIC) | Follow-up visits at 1, 2, 3, and 4 weeks after the IV ketamine infusion
  PGIC is a seven-point single-item scale ranging from 'very much worse' to 'very much improved' worse' with 'no change' as the mid-point that evaluates improvement with treatment during a clinical trial.
Periprocedural adverse effects | Baseline visit: During the infusion
  Variations of heart rate (beats per minute)
Periprocedural adverse effects | Baseline visit: During the infusion
  Variations of blood pressure (mmHg)
Periprocedural adverse effects | Baseline visit: During the infusion
  Variations of pulse oxygen saturation (percentage of hemoglobin carrying oxygen)
Periprocedural adverse effects | Baseline visit: During the infusion
  Presence of dizziness, nausea, chest pain, shortness of breast
Postprocedural adverse effects | Baseline visit: During 60-90 minutes after the procedure
  Variations of heart rate (beats per minute)
Postprocedural adverse effects | Baseline visit: During 60-90 minutes after the procedure
  Variations of blood pressure (mmHg)
Postprocedural adverse effects | Baseline visit: During 60-90 minutes after the procedure
  Variations of pulse oxygen saturation (percentage of hemoglobin carrying oxygen)
Postprocedural adverse effects | Baseline visit: During 60-90 minutes after the procedure
  Presence of dizziness, nausea, chest pain, shortness of breast

CONTACTS AND LOCATIONS:
Overall Officials: Igor Wilderman, MD, Principal Investigator — Wilderman Medical Clinic
Locations (1):
- Wilderman Medical Clinic, Thornhill, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will be available according to reasonable demands.